CLINICAL TRIAL: NCT05289817
Title: Effectiveness of Transcutaneous Electrical Stimulation on the Autonomous and Cardiovascular System on Healthy Young People; a Prospective, Randomized, Single-blind, Controlled Pilot Study
Brief Title: Effects of Transcutaneous Electrical Stimulation on the Autonomous Nerve System in Healthy Young People
Acronym: ESautonomous
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Alicia Martínez Rodríguez, Lecturer, PhD, MSC, PT. Faculty of Physical Therapy., Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/011
Record Dates: First submitted 2022-02-10; First posted 2022-03-21 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers; Cardiovascular System; Autonomic Nervous System
Keywords: Electric Stimulation Therapy; Transcutaneous Electric Nerve Stimulation; Parasympathetic Nervous System; Stellate Ganglion; Hearth Rate; Blood Pressure

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized, three-armed, sham-controlled, single-blind, exploratory clinical trial in healthy subjects
Who Masked: Participant
Masking Description: Allocation concealment, stratified by sex, will be ensured by the use of sealed envelopes containing the treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcutaneous Vagus Electrical Nerve Stimulation (t-VNS) (Experimental): Transcutaneous electrical stimulation will be delivered by trains for twenty minutes to the right cymba conchae at the ear.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation (t-VNS)
- Transcutaneous Sympathetic Ganglion Electrical Nerve Stimulation (t-SNS) (Active Comparator): Transcutaneous electrical stimulation will be delivered continuously for twenty minutes to the cervicothoracic region.
  Interventions: Device: Transcutaneous Sympathetic Ganglion Electrical Stimulation (t-SES)
- Sham Transcutaneous Vagus Electrical Nerve stimulation (sham t-VNS) (Sham Comparator): Transcutaneous electrical stimulation will be delivered by trains for twenty minutes to the right scapha at the ear.
  Interventions: Device: Sham Transcutaneous vagus nerve stimulation (Sham t-VNS)

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation (t-VNS) — Type of device and current: portable machine, low frequency current, constant current Type of wave: square biphasic pulses Pulse duration: 350 microseconds Frequency: 10 Hz Number of channels: one Location and electrodes: cymba conchae at right ear (vagus branch nerve area); a clip electrode will be applied with its cathode on anterior cymba conchae, the anode placed behind.
  Amplitude: from 2 times the perception threshold (individualized) at a comfortable, non-painful amplitude, and to a maximum of 9 mA. It will be increased, if necessary, each 5 minutes in order to maintain the same level of tingling sensation On-Off times: trains of 30 s on, 5 s rump up, 1 s rump down, 24 s off Duration: 20 minutes
  Arms: Transcutaneous Vagus Electrical Nerve Stimulation (t-VNS)
Device: Transcutaneous Sympathetic Ganglion Electrical Stimulation (t-SES) — Type of device and current: portable machine, low frequency current, constant current Type of wave: square biphasic pulses Pulse duration: 350 microseconds Frequency: 5 Hz Number of channels: two Location and electrodes: cervicothoracic area (stellate ganglion region); first channel: new 5 cm x 5 cm self-adhesive electrodes will be applied at 1-1.5 cm both sides of the vertebral spinous processes, approximately from C7 to T4, upper cathode on the left side of C7 and lower cathode on the right side.
  Amplitude: 2 mA above the muscle contraction threshold (individualized) at a comfortable, non-painful amplitude and to a maximum of 25 mA. It will be increased, if necessary, each 5 minutes in order to maintain the same level of muscle contraction On-Off times: no trains, continuously delivered Duration: 20 minutes
  Arms: Transcutaneous Sympathetic Ganglion Electrical Nerve Stimulation (t-SNS)
Device: Sham Transcutaneous vagus nerve stimulation (Sham t-VNS) — Type of device and current: portable machine, low frequency current, constant current Type of wave: square biphasic pulses Pulse duration: 350 microseconds Frequency: 10 Hz Number of channels: one Location and electrodes: scapha at right ear (non vagus innervated region); a clip electrode will be applied with its cathode on anterior scapha, the anode placed behind.
  Amplitude: from 2 times above the perception threshold (individualized) at a comfortable, non-painful amplitude, and to a maximum of 9 mA. It will be increased, if necessary, each 5 minutes in order to maintain the same level of tingling sensation On-Off times: trains of 30 s on, 5 s rump up, 1 s rump down, 24 s off Duration: 20 minutes
  Arms: Sham Transcutaneous Vagus Electrical Nerve stimulation (sham t-VNS)

SUMMARY:
Cardiovascular disease is one of the most important causes of death and disability in the world. An autonomic imbalance is associated to cardiovascular risks and disorders. Electrical stimulation (ES) applied by surface electrodes is a non-invasive therapeutic approach with low side-effects. In the last years, some studies had investigated the effects of ES on the autonomic nervous system and cardiovascular system. However, different intensities, frequencies and electrode locations had been used, which makes difficult to clarify the optimal parameters.

The aim of this study is to analyze the effects of ES on autonomic nervous modulation in healthy subjects comparing three different locations of application for ES.

Participants will be aleatory assigned to one of three groups for a single-session of 20-minute transcutaneous ES: a) an auricular intermittent ES in an area that is believed to be connected to the vagal nerve (cymba conchae); b) an auricular sham intermittent ES, meaning a real ES but applied on an ear location not connected to the vagal nerve (scapha); and c) an upper back continuous ES (C7-T4), a placement that is thought to be connected to the stellate (sympathetic) ganglion. All the protocols will be stated at a non-painful intensity. After that, the hand grip exercise will be executed.

The heart rate variability (HRV) and heart frequency (HR) will be measured in four main times: the baseline, in the final minutes of the ES, after the ES and after finishing the hand grip exercise. Blood pressure will be measured also at all the time points except during the ES due to the possibility of interferences. Adverse effects will be assessed after ES and 48 h later. The study will provide initial knowledge about how different electrical stimulation locations contribute to reduce sympathetic excitation and improve the sympathovagal balance.

DETAILED DESCRIPTION:
Electrical stimulation (ES) of the nervous system, also denominated as neuromodulation, has been investigated for diverse conditions as cardiovascular diseases, chronic pain and psychiatric conditions. It is unknown which locations and parameters can be more effective and better tolerated. The transcutaneous ES is a non-invasive technique which has fewer side-effects than subcutaneous vagus nerve stimulation.

The aim of this study is to analyze the acute effects of transcutaneous ES on autonomic nervous modulation by heart rate variability (HRV), heart frequency (HF) and blood pressure (BP) in healthy subjects comparing three different locations for the ES, before and after a hand-grip exercise. In addition, the tolerance to the current, the side-effects and the perceived exertion will be compared.

Once the participants have given their informed consent and had been checked for exclusion criteria, are invited to an experimental session. Subjects will be advised to refrain from caffeine or alcohol for 12 h and vigorous exercise for at least 24h prior to the intervention.

The participants will remain sitting during the entire session and will be instructed to stay awake and avoid movement. Grip strength will be evaluated by a hydraulic dynamometer (Saehan model SH5001). Participants will remain seated on a chair with their feet and trunk supported, shoulders adducted, elbows flexed at 90º, forearms in neutral position, and wrists with 0º-30º extension. Subjects will be instructed to perform a maximum isometric contraction for three to five seconds, and the peak force will be recorded. Three evaluations will be made with an interval of one minute between them. If the examiner would recognize some compensatory movement by the participant, a new measurement would be taken and registered.

The volunteers will be randomized by sex to one of three groups: cymba conchae at the right ear (active group); C7-T4 placement (active group), scapha at the right ear (sham-group). These three arms will be denominated as Transcutaneous Vagus Electrical Nerve Stimulation (t-VNS); Transcutaneous Sympathetic Ganglion Electrical Nerve Stimulation (t-SNS); and Sham Transcutaneous Vagus Electrical Nerve Stimulation (sham t-VNS), and. Allocation concealment, stratified by sex, will be ensured by the use of sealed envelopes containing the treatment allocation. The sequence will be generated using a computer program by a researcher not implicated in the experimental sessions. The envelopes will be opened just before determining the amplitude for stimulation. The stimulation location will be wiped down with alcohol and the minimum intensity, at which the stimulus is perceived, will be evaluated for the auricular locations, whereas minimum amplitude for muscle contraction between the electrodes will be assessed in cervico-thoracic location.

After 15 minutes of resting, the first assessment (baseline) will be taken (HRV, HR and blood pressure) for 5 minutes. The respiratory frequency will be checked every 5 minutes.

Then the randomized ES will be applied for 20 minutes using the same TENSMED S82 (Enraf Nonius, The Netherlands) symmetrical and rectangular biphasic pulses, at 350 microseconds of phase duration. It will be applied at 10 Hz (t-VNS and sham t-VNS) or 5 Hz (t-SNS). Both the two protocols applied to the auricular region (t-VNS and sham t-VNS) will be delivered by trains, whereas a continuous ES will be selected for the (t-SNS). The minimum amplitude for auricular stimulations (t-VNS and sham t-VNS) will be twice the perception threshold, at a comfortable intensity under the discomfort threshold (pain onset). It will be increased during the stimulation only if the sensation is clearly decreased to a maximum of 9 mA. The perception threshold will be set increasing amplitude by 0.5 mA each 3 seconds from 0 mA. Amplitude in t-SNS will be set at a muscle contraction at a comfortable intensity (under discomfort threshold or pain onset). The motor threshold will be determined by increasing amplitude 0.5 mA each 3 seconds from the perception threshold until a motor contraction is observed. The initial amplitude will be 2 mA over this threshold. It will be increased during the stimulation only if the stimulus falls down (to a maximum of 25 mA).

Another 5-minute period after ES will be recorded and then the 3-minute hand grip exercise (SH5001, Saehan, Korea) at 30% of maximum strength will be required.

The final assessment of cardiovascular and autonomous variables will be obtained during the last 15 minutes. The rating of perceived exertion will be asked (Borg-CR10) whereas a VAS (0 denoting no sensation at all; 10 = indicating discomfort or pain onset) will be used to rate the tolerance to ES. The possible side-effects will be also checked.

The participants will be asked upon completion of the session their presumed group assignment.

Adverse effects will be checked again 48 h after finishing the experimental session.

The ES and the acquisition of the data will be done by physical therapists, but analysis of the main variables will be done by a cardiologist with the assistance of one of the physical therapists with specific knowledge in the area. The data will be introduced by a third researcher, and accuracy of the data will be checked selecting 50% of the data from each arm, by random software. If some mistakes will emerge, then the complete check will be done. The traditional statistical analysis will be reinforced by Bayesian inferences.

This is a pilot study. The objective is to check if there are statistically significant effects from the stimulation on the variables: cardiac variability, heart rate and blood pressure, before or after an isometric exercise of pressure.

For the comparison of the results obtained in the three groups of subjects, the analysis of variance or rank test procedures will be used, based on the normality or non-normality of the data obtained.

The effect of time will be assessed through a longitudinal data analysis that takes into account the dependence. For this purpose, the repeated measures Anova or Friedman's test will be used, in the parametric or non-parametric assumption, as a global comparison procedure. Possible interactions and dependence relationships between measured variables and time will be studied by means of linear regression analysis, generalised linear and/or generalised kernel-type non-parametric modelling.

Comparisons between groups (Anova or its non-parametric equivalent) will be complemented by means of their equivalents in Bayesian analysis, in order to reinforce the information provided by the p-values obtained in each procedure. For this purpose, the corresponding Bayes factors (Kass and Raftery, 1995) and the posteriori distributions of the estimated parameters will be calculated, thus increasing the precision of the confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* University students and academic or administrative staff, non smokers, self-perceived as healthy

Exclusion Criteria:

* No history of neurological, neurosurgical, psychiatric, cardiological disease, pulmonary disease, syncope, seizure, head trauma, cranial or neck surgery, aneurisms, or any condition or treatment which could affect the functioning of the autonomous nerve system or the cardiovascular system (by self-report).
* BMI of 30 or over
* High blood pressure (systolic blood pressure of 140 mmHg or over, or diastolic blood pressure of 90 mmHg or over)
* Spontaneous respiratory rate under 10 breaths per minute
* Professional athletes
* Inability to reach the minimum amplitude required during electrical stimulation
* Any arm or hand pain (dominant side)
* Any contraindication for electrical stimulation (pregnancy or risk or being pregnant, any implanted electronical device, irritation or pain at the skin location for the electrodes, intolerance to electrical stimulation) or any condition which could affect the placement of the electrodes or the perception of the electrical stimulus.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
RR | 5 minutes before Electrical Stimulation, During 20 minutes Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  The time of RR intervals (ms) will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland). The mean values of RR intervals (ms) and the standard deviation of all RR intervals (ms) will be obtained.
RMSSD | 5 minutes before Electrical Stimulation, During 20 minutes Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  Root mean square of successive RR interval differences (ms). It will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland).
pNN50 | 5 minutes before Electrical Stimulation, During 20 minutes Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  Relative number of successive RR interval pairs that differ more than 50 ms (percentage). It will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland).
HF | 5 minutes before Electrical Stimulation, During 20 minutes Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  High frequency refers to HRV frequency band (0.15-0.4 Hz). It will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland).
LF | 5 minutes before Electrical Stimulation, During 20 minutes Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  Low frequency refers to HRV frequency band (0.04-0.15 Hz). It will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland).
LF/HF | 5 minutes before Electrical Stimulation, During 20 minutes Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  The ratio of LF to HF power will be calculated along with normalised LF/HF where baseline values will set to 1. It will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland).
SD1 | 5 minutes before Electrical Stimulation, During 20 minutes Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  The poincaré plot short term variability (ms). It will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland).
SD2 | 5 minutes before Electrical Stimulation, During 20 minutes Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  The poincaré plot long term variability (ms). It will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland).
SD2/SD1 | 5 minutes before Electrical Stimulation, During 20 minutes Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  Poincaré plot long and short term variability ratio. It will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland).
Mean heart rate | 5 minutes before Electrical Stimulation, during 20 minutes of Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  The mean frequency will be obtained from Polar S800 with Polar T31 transmitter (Polar Electro, Kempele, Finland), and it will be extracted with Kubios software (University of Eastern Finland, Kuopio, Finland).
Systolic blood pressure | 5 minutes before Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  Blood pressure will be continuously acquired by SOMNOtouch NIBP (Somnomedics, GmbH, Randersacker, Germany) that is an ambulatory cuffless device for continuous (beat-to-beat), noninvasive BP monitoring. The system consists of a finger photoplethysmograph and three ECG leads, connected to a watch-like control unit placed at the wrist level and equipped with a screen where beat-to-beat pulse waveform, ECG, and PTT changes are displayed. All these measurements are unified to obtain systolic blood pressure in mmHg.
Diastolic blood pressure | 5 minutes before Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  Blood pressure will be continuously acquired by SOMNOtouch NIBP (Somnomedics, GmbH, Randersacker, Germany) that is an ambulatory cuffless device for continuous (beat-to-beat), noninvasive BP monitoring. The system consists of a finger photoplethysmograph and three ECG leads, connected to a watch-like control unit placed at the wrist level and equipped with a screen where beat-to-beat pulse waveform, ECG, and PTT changes are displayed. All these measurements are unified to obtain the diastolic blood pressure in mmHg.
Mean arterial pressure | 5 minutes before Electrical Stimulation, 5 minutes after Electrical Stimulation, During 3 minutes hand-grip exercise, 15 minutes after hand grip exercise
  Blood pressure will be continuously acquired by SOMNOtouch NIBP (Somnomedics, GmbH, Randersacker, Germany) that is an ambulatory cuffless device for continuous (beat-to-beat), noninvasive BP monitoring. The system consists of a finger photoplethysmograph and three ECG leads, connected to a watch-like control unit placed at the wrist level and equipped with a screen where beat-to-beat pulse waveform, ECG, and PTT changes are displayed. All these measurements are unified to obtain the mean arterial pressure in mmHg.

SECONDARY OUTCOMES:
Electrical simulation tolerance | 20 minutes after initiating electrical stimulation
  The participants will be asked to rate their feelings during electrical stimulation by placing a solid vertical line on a 100-mm scale anchored by opposing descriptors (0=no sensation at all; 100 = pain onset or discomfort). Visual Analogue Scale (VAS) will be "scored" by measuring the rating with a ruler (millimeters)
Rating of perceived effort | Immediately after the hand grip exercise
  Subjective feelings of effort and fatigue of the arm using de Borg CR-10, from 0 (nothing at all) to 10 (almost maximal)
Adverse effects | At 20 minutes after initiating electrical stimulation and at 48 hours after the electrical stimulation
  All posible adverse effects due to the electrical stimulation and the electrodes will be checked by a questionnaire

OTHER OUTCOMES:
Blind outcome assessment | 15 minutes after the hand grip exercise
  Subjects will be asked to tell if they think they were assigned to an active or a sham group
Amplitude of electrical stimulation | 20 minutes of electrical stimulation
  mA are recorded every 5 minutes; mean mA is obtained by adding amplitude used in each 5 minutes period divided by 4, as 20 minutes is the total duration of the electrical stimulation
Respiratory frate | 5 minutes before Electrical Stimulation, during 20 minutes of Electrical Stimulation, 5 minutes after Electrical Stimulation, 15 minutes after hand grip exercise
  Number of breaths over the course of one minute. It will be visually monitored each 5 minutes, except during the grip exercise
Body Mass Index | Baseline
  Body Mass Index (kg/m^2)
Somatotype | Baseline
  Height (cm); Weight (Kg); Skinfolds (mm); Biepicondylar breadth of the humerus and femur (cm); Upper arm, elbow flexed and tensed, calf girth (cm).
  Sheldon's somatotype classification is computed using the following equations:
  Endomorphy = -0,7182 + 0,1451X - 0,00068X^2 + 0,0000014X^3 where: X= sum of skinfolds (triceps + subscapular + supraspinale)*170.18 / Height
  Mesomorphy= (0.858*Biepicondylar breadth of the humerus + 0,601*Biepycondilar breadth of the femur + 0.188*Corrected Arm girth + 0.161*Corrected Calf girth) - (Height*0.131) + 4.5.
  Ectomorphy = Height - Weight ratio (HWR) according to the following conditions:
  1. If HWR≥40.75, then: Ectomorphy = HWR×0.732-28.58
  2. If HWR<40.75 but >38.25, then: Ectomorphy = HWR×0.463-17.63
  3. If HWR≤38.25, then: then: Ectomorphy = 0.1
Waist and hip circumferences | Baseline
  Cm of waist circumference and hip circumference. The waist-to-hip ratio will be calculated by dividing waist circumference by hip circumference.
Waist to hip ratio | Baseline
  It will be calculated by dividing waist circumference by hip circumference
Body composition (bio impedance) | Baseline
  percentage of fat, muscle, water and bone (bio impedance)
Body density (BD) | Baseline
  BD=1.0988-0.0004*(skinfolds in mm of triceps + subscapular +biceps+ supraspinale +abdominal+ front thigh +medial calf)
Percent body fat (percentage BF) from body density (BD) | Baseline
  Percentage BF from BD = (4.570/BD-4.142) *100.
Fat mass | Baseline
  Fat mass (Kg) = body weight (kg) * percentage body fat/100
Fat-free mass | Baseline
  Fat-free mass (Kg) = body weight (kg)-fat mass (kg)
Fat mass index (FMI) | Baseline
  FMI is calculated by dividing the fat mass by the stature-squared: fat mass/height^2
Fat-free mass index (FFMI) | Baseline
  FFMI is calculated by dividing the fat-free mass by the stature-squared: fat-free mass/height^2
Short International Physical Activity questionnaire (IPAQ) | Baseline
  IPAQ assesses physical activity as walking, moderate-intensity activities and vigorous intensity activities; frequency (days per week) and duration (time per day) are collected separately for each specific type of activity. Computation of the total score requires summation of the duration (in minutes) and frequency (days) of each type of activity. Another measure is computed by weighting each type of activity by its energy requirements defined in METS (multiples of the resting metabolic rate) to yield a score in MET-minutes. These following values are used for the analysis of IPAQ data: Walking = 3.3 METs, Moderate PA = 4.0 METs and Vigorous PA = 8.0 METs. The higher the MET-minutes the more intense the physical activity is, with 0 indicating no activity at all. As there are no established thresholds for presenting MET-minutes, the IPAQ Research Committee proposes that these data are reported as comparisons of median values and interquartile ranges for different populations.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Martínez-Rodríguez, PhD, Principal Investigator — Universidade da Coruña (UDC)
Locations (1):
- Universidade da Coruna, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No